CLINICAL TRIAL: NCT01195207
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Intravenous Study in Healthy Subjects and a Multiple-Dose Intravenous Study in Asthmatic Subjects to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of CNTO 3157
Brief Title: A Phase 1 Study of CNTO 3157 in Healthy Volunteers and Patients With Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centocor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CR017095
Record Dates: First submitted 2010-09-02; First posted 2010-09-06 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Asthma
Keywords: CNTO 3157; healthy volunteers; asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (8):
- 001 (Experimental): CNTO 3157 or placebo 0.003 mg/kg CNTO 3157 or placebo infusion
  Interventions: Biological: CNTO 3157 or placebo
- 002 (Experimental): CNTO 3157 or placebo 0.01 mg/kg CNTO 3157 or placebo infusion
  Interventions: Biological: CNTO 3157 or placebo
- 003 (Experimental): CNTO 3157 or placebo 0.03 mg/kg CNTO 3157 or placebo infusion
  Interventions: Biological: CNTO 3157 or placebo
- 004 (Experimental): CNTO 3157 or placebo 0.1 mg/kg CNTO 3157 or placebo infusion
  Interventions: Biological: CNTO 3157 or placebo
- 005 (Experimental): CNTO 3157 or placebo 0.3 mg/kg CNTO 3157 or placebo infusion
  Interventions: Biological: CNTO 3157 or placebo
- 006 (Experimental): CNTO 3157 or placebo 1 mg/kg CNTO 3157 or placebo infusion
  Interventions: Biological: CNTO 3157 or placebo
- 007 (Experimental): CNTO 3157 or placebo 3 mg/kg CNTO 3157 or placebo infusion
  Interventions: Biological: CNTO 3157 or placebo
- 008 (Experimental): CNTO 3157 or placebo 10 mg/kg CNTO 3157 or placebo infusion
  Interventions: Biological: CNTO 3157 or placebo

INTERVENTIONS:
Biological: CNTO 3157 or placebo — 0.003 mg/kg CNTO 3157 or placebo infusion
  Arms: 001
Biological: CNTO 3157 or placebo — 0.03 mg/kg CNTO 3157 or placebo infusion
  Arms: 003
Biological: CNTO 3157 or placebo — 10 mg/kg CNTO 3157 or placebo infusion
  Arms: 008
Biological: CNTO 3157 or placebo — 0.01 mg/kg CNTO 3157 or placebo infusion
  Arms: 002
Biological: CNTO 3157 or placebo — 1 mg/kg CNTO 3157 or placebo infusion
  Arms: 006
Biological: CNTO 3157 or placebo — 3 mg/kg CNTO 3157 or placebo infusion
  Arms: 007
Biological: CNTO 3157 or placebo — 0.3 mg/kg CNTO 3157 or placebo infusion
  Arms: 005
Biological: CNTO 3157 or placebo — 0.1 mg/kg CNTO 3157 or placebo infusion
  Arms: 004

SUMMARY:
This is a phase 1, safety study of CNTO 3157 in healthy subjects and subjects with asthma.

DETAILED DESCRIPTION:
A phase 1, randomized (study drug assigned by chance), double blind (neither physician nor patient knows if CNTO 3157 or placebo has been assigned), placebo controlled, single, ascending-dose study of CNTO 3157 in healthy volunteers and multiple dose study in patients with asthma. This study will compare the effects (both good and bad) of CNTO 3157 to those of placebo. The purpose of this study is to evaluate the safety and potential side effects of CNTO 3157 given to healthy volunteers and patients with asthma. In addition, the investigators will measure how much study drug is in the blood following a dose of CNTO 3157, and determine if the body makes antibodies to it. (An antibody is a protein made by the body in response to a foreign substance). Safety assessments will be performed throughout the study and include obtaining and evaluating laboratory tests, vital signs (e.g., blood pressure), and the occurrence and severity of adverse events. There will be 2 parts to this study. The first part of this study will involve healthy volunteers, and the second part of the study will involve patients with asthma. About 56 healthy volunteers and 16 asthmatic patients will take part. Volunteers will be required to stay at the research center after study agent administration for an inpatient portion of the study and then return for required out-patient visits. Up to approximately 8 different dose levels will be studied. CNTO 3157 will be administered by IV infusion. The duration of volunteer participation will be up to 21 weeks in Part 1 and up to 24 weeks in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female between 18 and 55 years of age inclusive with no clinically significant abnormalities and have a body weight of 50 to 100 kg
* Patients with asthma must have been diagnosed at least 6 months prior to participation in the study

Exclusion Criteria:

* Currently have or have a history of any clinically significant medical illness or medical disorders the investigator considers should exclude the subject, including (but not limited to) cardiovascular disease, neuromuscular, hematological disease, immune deficiency state, respiratory disease (other than asthma for Part 2), hepatic or GI disease, neurological or psychiatric disease, ophthalmological disorders, neoplastic disease, renal or urinary tract diseases, or dermatological disease
* Have a positive pregnancy test at screening or prior to dose administration
* Have smoked tobacco or related products within 6 months prior to dosing
* Donated blood equal to or greater than ¿450 mL within 60 days prior to participation in the study
* Recent history (within previous 6 months) of alcohol or drug abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2010-06; Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of CNTO 3157 by evaluating laboratory tests, vital signs (e.g., blood pressure), and the occurrence and severity of adverse events | Week 21 for Part 1 and Week 24 for Part 2

SECONDARY OUTCOMES:
Evaluate the effects of CNTO3157 on the body and the effects of the body on CNTO 3157 (Pharmacokinetics (PK), Pharmacodynamics (PD)) | Week 21 for Part 1 and Week 24 for Part 2
Immune response (Immunogenicity) | Week 21 for Part 1 and Week 24 for Part 2
Clinical Response | Week 21 for Part 1 and Week 24 for Part 2

CONTACTS AND LOCATIONS:
Overall Officials: Centocor, Inc. Clinical Trial, Study Director — Centocor, Inc.
Locations (4):
- Belgium (2):
  - Antwerp
  - Merksem
- Berlin, Germany
- Harrow, United Kingdom